CLINICAL TRIAL: NCT07116577
Title: A Single-Arm, Exploratory Study of Palliative Radiotherapy Combined With Iparomlimab and Tuvonralimab, Trifluridine/Tipiracil (TAS-102), and Bevacizumab in Later-Line Treatment of Advanced Colorectal Cancer
Brief Title: Radiotherapy Combined QL1706, TAS-102 and Bevacizumab in mCRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinan Central Hospital (Other)
Responsible Party: Principal Investigator, Meili Sun, Director of Department of Oncology, Jinan Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250710004
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: mCRC
MeSH Terms: interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Palliative radiotherapy combined with iparomlimab and tuvonralimab (QL1706), trifluridine/tipiracil (TAS-102), and bevacizumab.
  Interventions: Radiation: Palliative radiotherapy; Drug: Iparomlimab and tuvonralimab; Drug: TAS-102; Drug: Bevacizumab

INTERVENTIONS:
Radiation: Palliative radiotherapy — Conventional fractionation, low-dose hypofractionated radiotherapy, or high-dose hypofractionated radiotherapy may be employed.
Drug: Iparomlimab and tuvonralimab — 5 mg/kg, intravenously infused on Day 1 of each cycle, administered every 3 weeks (with each cycle defined as 21 days).
Drug: TAS-102 — 35 mg/m², orally twice daily on Days 1 to 5 and Days 8 to 12 of each cycle, with each cycle spanning 28 days (4 weeks).
Drug: Bevacizumab — 7.5 mg/kg via intravenous infusion on Day 1 of each 21-day cycle.

SUMMARY:
This single-center, single-arm, prospective study plans to enroll patients with advanced colorectal cancer who have failed first-line or higher systemic therapies. Participants will receive a combination of iparomlimab and tuvonralimab (QL1706), trifluridine/tipiracil (TAS-102), bevacizumab, and palliative radiotherapy. The efficacy and safety of this combination therapy will be evaluated by assessing objective response rate (ORR), progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years .
* Histologically confirmed unresectable colorectal adenocarcinoma.
* Patients must have received at least one prior line of oxaliplatin-, irinotecan-, or 5-FU-based therapy with documented progression or intolerance.
* Documented KRAS and BRAF mutation status (mutant or wild-type) must be available.
* Palliative radiotherapy targeting primary or metastatic lesions is planned.
* At least one measurable lesion per RECIST v1.1 exists.
* ECOG score of 0-1 and life expectancy ≥12 weeks.
* Adequate bone marrow, hepatic, and renal function must be demonstrated.
* Fertile patients commit to using effective contraception during and for 6 months post-treatment.

Exclusion Criteria:

* History of Grade ≥3 immune-related adverse events (irAEs) from prior immunotherapy deemed contraindications for retreatment.
* Radiation or systemic anticancer therapy within 14 days prior to first study treatment.
* Active CNS metastases and/or leptomeningeal disease (LMD). Symptomatic interstitial lung disease (ILD), active pneumonitis, uncontrolled infections, or non-healing wounds/fistulae.
* Intestinal perforation risks: active diverticulitis, intra-abdominal abscess, GI obstruction, or cancer-related peritoneal carcinomatosis.
* Uncontrolled or symptomatic serous cavity effusions (pleural, ascites, pericardial).
* Uncontrolled cardiovascular/cerebrovascular diseases.
* Medical/social conditions that may compromise study results or lead to premature termination per investigator judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | approximately 4 months after the last subject participating in
  The time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
PFS | approximately 12 months after the last subject participating in
  the proportion of subjects with complete response (CR) and partial response (PR) according RESIST1.1 in total subjects.
OS | approximately 12 months after the last subject participating in
  The time from the starting date of study drug to the date of death due to any cause.
DCR | approximately 4 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease(SD) in total subjects
Safety (adverse event) | Up to approximately 2 years.
  The rates of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Meili Sun, Director, Department of Oncology, MD, PhD,, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China